CLINICAL TRIAL: NCT01750112
Title: An Open Non Comparative Multicenter Prospective Study to Evaluate Efficacy and Safety of Macrolane VRF20 in Treatment of Pectus Excavatum
Brief Title: Treatment of Pectus Excavatum Deformity Using Macrolane Filler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Collaborators: Pharma Consulting Group AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31GC1201
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2017-05

CONDITIONS: Pectus Excavatum Deformity
Keywords: Pectus excavatum; funnel chest; sunken chest
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macrolane VRF20 (Experimental): All subjects will receive treatment with Macrolane VRF20 to correct pectus excvatum deformity.
  Interventions: Device: Macrolane VRF20

INTERVENTIONS:
Device: Macrolane VRF20 — Injection treatment with Macrolane VRF20

SUMMARY:
This is a prospective, open, non-comparative and baseline-controlled study to evaluate efficacy and safety of Macrolane VRF20 treatment in 40 subjects with pectus excavatum deformity.

Each subject participating in the study will be treated with approximately 50-150 ml of Macrolane VRF20. The amount of study product used will be individually determined in order to achieve an optimal correction of the deformity in each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Give verbal and written informed consent to participate in the study.
2. Be a healthy male of 18 years or more.
3. Have a pectus excavatum deformity without functional problems; score 4 in items 10, 11 and 12 of the PEEQ, indicating there is no functional impairment due to the pectus excavatum deformation.
4. Present normal cardiac function as assessed by ECG and echocardiogram.
5. Present normal pulmonary function as assessed by pulmonary function test.
6. Present a chest X-ray taken within 12 months prior to the baseline visit, without clinically significant defects to heart, lungs, skeleton, ribs, sternum or spinal cord except for the pectus excavatum defect, in the opinion of the Investigator.
7. Have the ability to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Score 1, 2 or 3 in either of items 10, 11 and 12 of the PEEQ, indicative of functional problems due to the pectus excavatum deformity.
2. Previous treatment for the same indication.
3. Known or suspected hypersensitivity to hyaluronic acid based products.
4. BMI < 20.
5. A history of severe allergies manifested by a history of anaphylaxis, or a history or presence of multiple severe allergies (as judged by the Investigator).
6. Known allergy to any anesthesia planned during the study.
7. Presence of autoimmune disease or other chronic disease that in the opinion of the Investigator may interfere with the outcome of the study.
8. Subjects with bleeding disorders or subjects who are taking thrombolytics or anticoagulants, or have taken inhibitors of platelet aggregation, including non-steroidal anti-inflammatory agents and acetylsalicylic acid, two weeks before treatment.
9. Subjects on immunomodulatory therapy (suppressive or stimulatory).
10. Subjects with contraindications for MRI, such as presence of pacemaker, clips or splinter, or tendency for claustrophobia.
11. Any condition which in the opinion of the Investigator makes the subject unsuitable for inclusion (e.g., subjects not likely to participate for the duration of the study).
12. Use of any investigational drugs or devices within 30 days prior to baseline.
13. Subjects who are study site staff for this study, or close relatives of the study site staff, as well as subjects who are employed by the Sponsor company, or close relatives of employees at the Sponsor company.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-12; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
PEEQ | Jul 2016
  To evaluate improvement from baseline in general self-esteem and emotion at 1, 3, 6, 12 and 24 months after treatment with Macrolane VRF20, using a modified version of the pectus excavatum evaluation questionnaire (PEEQ) before and after treatment.
Subject satisfaction | Jul 2016
  Evaluate subject satisfaction at 1, 3, 6, 12 and 24 months after treatment.
Duration | Jul 2016
  Estimate duration of Macrolane VRF20 calculated using MRI images at 12 months (and 24 months for a subset of patients).
Placement | Jul 2016
  Assess placement using MRI at 1 and 12 months post treatment.
Adverse event | Jul 2016
  To study safety throughout the study period, i.e. up to 24 months after treatment, based on evaluation of reported Adverse Events.
Downtime | Jul 2016
  Evaluate recovery time after treatment using 14-days subject diary.
Downtime 2 | Jul 2016
  Evaluate days hospitalized or on sick leave after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Per Hedén, MD, PhD, Principal Investigator — Akademikliniken; Raphael Sinna, MD, PhD, Principal Investigator — University Hospital of Amiens
Locations (2):
- Raphael Sinna, Amiens, France
- Per Heden, Stockholm, Sweden